CLINICAL TRIAL: NCT06130553
Title: PRIMROSE: A Modular Phase I/IIa, Multi-centre, Dose Escalation, and Expansion Study of AZD3470, a MTA Cooperative PRMT5 Inhibitor, as Monotherapy and in Combination With Anticancer Agents in Patients With Advanced/Metastatic Solid Tumors That Are MTAP Deficient
Brief Title: A Study of AZD3470, a PRMT5 Inhibitor, in Patients With MTAP Deficient Advanced/Metastatic Solid Tumors
Acronym: PRIMROSE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9970C00001; 165618 (Registry Identifier: IND)
Record Dates: First submitted 2023-10-19; First posted 2023-11-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors That Are MTAP Deficient
Keywords: solid tumor; MTAP deficient

STUDY DESIGN:
Intervention Model Description: This is a FTiH (first time in human), modular Phase I/IIa, open-label, multi-centre study of AZD3470, in participants with MTAP deficient advanced/metastatic solid tumors. The study consists of individual modules, each evaluating safety and tolerability of AZD3470 dosed as a monotherapy and in combination with specific treatments. Module 1 describes AZD3470 monotherapy, and will have at least two parts. Part A will include the dose escalation cohorts. Part B will include the dose optimization and expansion cohorts.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD3470 Monotherapy (Experimental): Part A dose escalation and back-fill cohorts and Part B dose optimization and expansion cohorts of varying doses of AZD3470
  Interventions: Drug: AZD3470

INTERVENTIONS:
Drug: AZD3470 — AZD3470 is a novel, potent and selective, second-generation, MTAP-selective, inhibitor of PRMT5.

SUMMARY:
This is a first time in human (FTiH) Phase I/IIa, open-label, multi-centre study of AZD3470 in participants with advanced or metastatic solid tumors with MTAP deficiency. The study consists of several study modules, evaluating the safety, tolerability, pharmacokinetic (PK), pharmacodynamics, and preliminary efficacy of AZD3470 as monotherapy or in combination with other anti-cancer agents.

DETAILED DESCRIPTION:
This first time in human, open-label, multi-centre study of AZD3470 in participants with advanced or metastatic solid tumors with MTAP deficiency follows a modular design. Module 1 Part A will include the dose escalation cohorts. Part B will include the dose optimization and expansion cohorts. New modules for combination treatments may be added in the future based on emerging data.

ELIGIBILITY:
Principle Inclusion Criteria:

* Participant must be at least 18 years of age or the legal age of consent in the jurisdiction in which the study is taking place, at the time of signing the ICF.
* Willing to provide archival and/or baseline tumor sample to meet the minimum tissue requirement for central MTAP deficiency testing.
* Participants must have received and progressed, are refractory or are intolerant to standard therapy for the specific tumor type. All participants are required to have had at least one prior line of treatment in the recurrent or metastatic setting.
* MTAP deficient tumors defined as evidence of homozygous deletion of one or more exons of the MTAP gene in tumor tissue AND/OR loss of MTAP expression in the tumor tissue.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* A minimum life expectance of 12 weeks in the opinion of the Investigator.
* Participants must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Adequate organ and bone marrow reserve function.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Principle Exclusion Criteria:

* Spinal cord compression or symptomatic and unstable brain metastases or leptomeningeal disease or primary malignancies of the central nervous system.
* Allogeneic organ transplantation.
* Any significant laboratory finding or any severe and uncontrolled medical condition.
* Any of the following cardiac criteria:
* LVEF ≤ 50%
* prior or current cardiomyopathy
* clinically active cardiovascular disease, or a history of myocardial infarction within the last 6 months
* uncontrolled angina or acute coronary syndrome within 6 months
* severe valvular heart disease
* uncontrolled hypertension
* risk of brain perfusion problems. Stroke or transient ischemic attack in the last 6 months, undergone coronary artery bypass graft, angioplasty or vascular stent
* chronic heart failure
* factors that increase the risk of QTc prolongation or risk of arrhythmic events
* Mean resting QTcF > 470 msec or any clinically important abnormalities in rhythm
* Use of therapeutic anti-coagulation for treatment of acute thromboembolic events.
* Serologic active hepatitis B or C infection.
* Known to have tested positive for Human immunodeficiency virus (HIV).
* Confirmed or suspected ILD/pneumonitis or history of (non-infectious) ILD/pneumonitis that required oral or IV steroids or supplemental oxygen
* Active gastrointestinal disease or other condition that would interfere with oral therapy.
* History of another primary malignancy.
* Unresolved toxicities from prior anti-cancer therapy, except alopecia and neuropathy.
* Prior treatment with a protein arginine methyltransferase 5 (PRMT5) inhibitor .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From time of informed consent to 28 days post last dose of AZD3470
  Number of participants with AEs and SAEs
Incidence of dose-limiting toxicities (DLT) | From first dose of study treatment until the end of Cycle 1 (each cycle is 21 days)
  Incidence of dose-limiting toxicities (DLT) as determined by number of patients with at least 1 dose-limiting toxicity (DLT). DLT is defined as an AE (adverse event) or abnormal laboratory value that occurs during the DLT period (defined as 21 days after start of study intervention) that is assessed as unrelated to the disease, intercurrent illness, or concomitant medications and meets any DLT criteria defined in the clinical study protocol

SECONDARY OUTCOMES:
Radiological response assessed by the Investigator evaluated according to RECIST v1.1 - ORR (Objective Response Rate) | From date of first dose of AZD3470 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years).
  Proportion of participants who have a confirmed complete or partial radiological response as determined by the Investigator according to RECIST v1.1
Radiological response assessed by the Investigator evaluated according to RECIST v1.1 - DoR (Duration of Response) | From date of first dose of AZD3470 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years).
  DoR - the time from date of first documented objective response (which is subsequently confirmed) until date of documented disease progression per Tumor RECIST v1.1 as assessed by the Investigator at local site or death due to any cause.
Radiological response assessed by the Investigator evaluated according to RECIST v1.1 - Best percentage change in tumor size | From date of first dose of AZD3470 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years).
  Best percentage change from baseline in TL (target lesion) tumor size is based on the RECIST 1.1. TL measurements as assessed by the Investigator.
Radiological response assessed by the Investigator evaluated according to RECIST v1.1 - PFS (Progression Free Survival) | From date of first dose of AZD3470 up until progression, or the last evaluable assessment in the absence of progression (approximately 2 years).
  PFS - defined as time from date of first dose (nonrandomized study parts) or date of randomization (randomized study parts) until progression per RECIST v1.1 as assessed by the Investigator at local site, or death due to any cause.
Radiological response assessed by the Investigator evaluated according to RECIST v1.1 - DCR (Disease Control Rate) at 12 weeks | From date of first dose of AZD3470 up until progression, or the last evaluable assessment in the absence of progression (for each patient this is expected to be measured at 12 weeks).
  DCR at 12 weeks defined as the percentage of participants who have a confirmed CR (complete response) or PR (partial response) or who have SD (stable disease) per RECIST 1.1 as assessed by the Investigator at local site and derived from the raw tumor data for at least 11 weeks after date of first dose to allow for an early assessment within the assessment window.
Overall Survival (OS) | From date of first dose of AZD3470 up until the date of death due to any cause (approximately 2 years).
  Overall Survival (OS) - defined as time from date of first dose (nonrandomized study parts) or date of randomization (randomized study parts) until the date of death due to any cause.
Module 1 Endpoints Part A (Dose escalation) Measurement of PK parameters: AUC | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (Dose escalation) Measurement of PK parameters: Area under the concentration time curve (AUC).
Module 1 Endpoints Part A (Dose escalation) Measurement of PK parameters: C-max | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (Dose escalation) Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max).
Module 1 Endpoints Part A (Dose escalation) Measurement of PK parameters: half life | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (Dose escalation) Measurement of PK parameters: Terminal elimination half-life (t 1/2)
Module 1 Endpoints Part A (Dose escalation) Measurement of PK parameters: Ae (excreted in urine) | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (Dose escalation) Measurement of PK parameters: amount of AZD3470 excreted in urine (Ae).
Module 1 Endpoints Part A (Dose escalation) Measurement of PK parameters: Clr (renal clearance) | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (Dose escalation) Measurement of PK parameters: renal clearance (Clr).
Module 1 Endpoints Part A drug-drug interaction (DDI) - Measurement of PK parameters of Midazolam: Cmax | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (DDI)- Plasma geometric mean ratio (Maximum observed plasma concentration of the study drug (C-max)) of Midazolam evaluated with and without AZD3470
Module 1 Endpoints Part A (DDI) - Measurement of PK parameters of Midazolam: AUC | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (DDI) - Plasma geometric mean ratio (Area under the concentration time curve (AUC)) of Midazolam evaluated with and without AZD3470
Module 1 Endpoints Part A (DDI) - Measurement of PK parameters of Dextromethorphan: Cmax | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (DDI)- Plasma geometric mean ratio (Maximum observed plasma concentration of the study drug (C-max)) of Dextromethorphan evaluated with and without AZD3470
Module 1 Endpoints Part A (DDI) - Measurement of PK parameters of Dextromethorphan: AUC | At predefined intervals throughout the treatment period (for each patient this is expected to be measured up to approximately 4 weeks)
  Part A (DDI) - Plasma geometric mean ratio (Area under the concentration time curve (AUC)) of Dextromethorphan evaluated with and without AZD3470
Module 1 Endpoints Part A pharmacodynamic backfill cohorts - Measurement of SDMA in tumor. | From screening baseline timepoint to up to four weeks on treatment timepoint.
  Part A pharmacodynamic backfill- Percentage change from baseline tumor SDMA as measured by immunohistochemistry.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (8):
  - Research Site, San Francisco, California
  - Research Site, West Hollywood, California
  - Research Site, New Haven, Connecticut
  - Research Site, Baltimore, Maryland
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Fairfax, Virginia
- Research Site, Melbourne, Australia
- China (3):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Shanghai
- Research Site, Villejuif, France
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa
- Research Site, Amsterdam, Netherlands
- Research Site, Seoul, South Korea
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home